CLINICAL TRIAL: NCT02386384
Title: TNFα (Tumor Necrosis Factor Alpha) and MFG-E8 (Milk Fat Globule-Epidermal Growth Factor 8): Novel Biomarkers to Predict Implantation Failure
Brief Title: TNFα and MFG-E8: Novel Biomarkers to Predict Implantation Failure
Status: Completed | Type: Observational
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Silvina Bocca, Associate Professor, Eastern Virginia Medical School
Other Study IDs: 15-01-FB-0004
Record Dates: First submitted 2015-03-06; First posted 2015-03-11 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Infertility; Recurrent Pregnancy Loss
Keywords: pregnancy failure
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control: Normal fertile
- Implantation Failure: Failure to conceive
- Recurrent Pregnancy Loss: 2 or more unexplained miscarriages

SUMMARY:
Question: Can implantation failure (IF) be predicted prior to in vitro fertilization (IVF)? A pilot, non-interventional, clinical study Prospective, controlled, cohort study

DETAILED DESCRIPTION:
The investigators hypothesize that TNFα and MFG-E8 cooperatively maintain the integrity of the normal endometrium, and that in patients with IF or with recurrent pregnancy loss (RPL) of unexplained origin, excessive TNFα increases the maternal shedding of MFG-E8, disrupting the normal protective effect of this protein, resulting in damage of the endometrial epithelium and impairing trophoblast invasion. The investigators propose that these molecules can be measured in local tissue (endometrium) as well as in serum as a reflection of increased inflammation and can therefore be used as markers of implantation and its failure. The investigators hypothesis is that TNFα is up-regulated in serum of women with implantation defects (IF and RM of unexplained origin) and this causes perturbation of MFG-E8 secretion. These results will provide first evidence demonstrating endometrial dysfunctions resulting from over-expression of pro-inflammatory molecules. The release of significant quantities of these molecules into serum broadens the maternal-fetal interface beyond the uterus and into the maternal circulation. The characterization of these molecules is essential to better understand, not only their biological effects, but also their potential as prognostic and diagnostic biomarkers for detection of IF. More importantly, these molecules could be potential therapeutic targets (perhaps intrauterine infusion of MFG-E8 for tissue repair, and/or oral administration of TNFα antagonists) to improve implantation outcomes. Two recent studies have reported the successful therapeutic use of recombinant human MFG-E8 (rhMFG-E8) in animals: one was used to decrease intestinal injury after whole body radiation (Ajakaiye et al, 2012), and the other was to mitigate inflammation and tissue injury after hemorrhagic stroke (Wang et al, 2012). Also, TNFα inhibitors have been shown to significantly increase IVF outcome in infertile patients (Winger et al, 2009 and 2008). In summary, these two pivotal studies show promising clinical uses of rhMFG-E8 in tissue repair/remodeling by decreasing apoptosis, and provide basis for their use as candidates for further clinical development in reproductive health.

Objectives: Here, the investigators seek to delineate novel diagnostic methods with the ultimate long term goal of designing directed therapies to improve embryo implantation competence.

* The specific aim is to quantify and correlate MFG-E8 and TNFα in serum and in endometrial biopsies of women in 3 groups: controls, IF and RM.
* The ultimate goal of this study is to provide data leading to a simple and quick test to measure soluble serum markers of IF/RM in order to discriminate prospectively between these groups of patients.
* To translate these findings into the use of modulators of these inflammatory molecules to improve pregnancy rates in patients with predicted implantation defects. It is widely known that "classic" markers of endometrial receptivity such as those provided by an invasive endometrial biopsy (with Hematoxilin-Eosin staining, or immuhistochemistry, or even with microarray technology) are not reliable to establish clear-cut diagnosis due to cycle-to-cycle variations and overlap of results.

ELIGIBILITY:
Inclusion Criteria:

* women 21-35y
* with no contraindication to pregnancy
* on no hormonal contraception
* normal uterine cavity
* absence of hydrosalpinges
* normal ovarian reserve (FSH<13 mIU/.ml or AMH>1 ng/ml or normal antral follicular count>10 total follicles <10 mm in diameter, American Society for Reproductive Medicine-ASRM 2012).
* Three groups of patients will be enrolled: 10 fertile controls (C1-10: women who are participating in the donor egg program as egg donors), 10 with unexplained implantation failure (IF1-10: patients who have failed IVF cycles -failure of implantation following 2 or more cycles with transfer of embryos of good quality-at least 2 cleaving embryos with 6-8 cells, grades 1- 3 (scale 1-highest and 5-poorest morphology score), and normal uterus, and 10 with recurrent unexplained first trimester miscarriages (RM1-10: 2 consecutive miscarriages under 10 weeks, after spontaneous or IVF conceptions).

Exclusion Criteria:

* contraindication to pregnancy
* use of hormonal contraception
* abnormal uterine cavity
* hydrosalpinges
* abnormal karyotype.
* women who are pregnant or planning to get pregnant in the cycle in which they are participating in this study
* women who have had a hysterectomy (previous removal of your uterus)
* have a current medical condition, which, in the opinion of the investigator, would result in hazards to the subject, should she participate in the study or have a current medical condition which would potentially confound the study results.

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women 21-35 years old attending an infertility clinic in an academic center
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
concentration of MFG-E8 and TNFα in serum and in endometrial biopsies controls, IF and RM. | 1 menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Silvina M Bocca, MD, PhD, Principal Investigator — Eastern Virginia Medical School

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu L, Anderson S, Oehninger S, Bocca S. Tumor necrosis factor alpha up-regulates endometrial milk fat globule-epidermal growth factor 8 protein production via nuclear factor kappaB activation, resulting in cell migration of epithelial cells. Fertil Steril. 2014 Feb;101(2):552-9. doi: 10.1016/j.fertnstert.2013.10.032. Epub 2013 Nov 18. PMID 24262600
- [Background] Schmitz C, Yu L, Bocca S, Anderson S, Cunha-Filho JS, Rhavi BS, Oehninger S. Role for the endometrial epithelial protein MFG-E8 and its receptor integrin alphavbeta3 in human implantation: results of an in vitro trophoblast attachment study using established human cell lines. Fertil Steril. 2014 Mar;101(3):874-82. doi: 10.1016/j.fertnstert.2013.12.015. Epub 2014 Jan 11. PMID 24424369
- [Background] Sarhan et al, MFG-E8 (milk fat globule EGF factor 8 protein) is a novel endometrial epithelial glycoprotein regulated by human chorionic gonadotropin (hCG) and secreted via microparticles. J Cell Signaling and Trafficking 2013
- [Background] Bocca SM, Anderson S, Amaker B, Swanson RJ, Franchi A, Lattanzio F, Oehninger S. Milk fat globule epidermal growth factor 8 (MFG-E8): a novel protein in the mammalian endometrium with putative roles in implantation and placentation. Placenta. 2012 Oct;33(10):795-802. doi: 10.1016/j.placenta.2012.06.015. Epub 2012 Jul 5. PMID 22770563
- [Background] Riggs RM, Bocca S, Anderson S, Franchi A, Rhavi BS, Oehninger S. Epithelial cell protein milk fat globule-epidermal growth factor 8 and human chorionic gonadotropin regulate stromal cell apoptosis in the human endometrium. Fertil Steril. 2012 Dec;98(6):1549-56.e3. doi: 10.1016/j.fertnstert.2012.07.1127. Epub 2012 Aug 24. PMID 22921913
- [Background] Franchi A, Bocca S, Anderson S, Riggs R, Oehninger S. Expression of milk fat globule EGF-factor 8 (MFG-E8) mRNA and protein in the human endometrium and its regulation by prolactin. Mol Hum Reprod. 2011 Jun;17(6):360-71. doi: 10.1093/molehr/gaq102. Epub 2010 Dec 21. PMID 21177637
- [Background] Bocca et al. Milk fat globule epithelial growth factor 8 (MFG-E8) regulates human endometrial endothelial cell adhesion and proliferation. Fertil Steril 2010, P423.
- [Background] Franchi A, Zaret J, Zhang X, Bocca S, Oehninger S. Expression of immunomodulatory genes, their protein products and specific ligands/receptors during the window of implantation in the human endometrium. Mol Hum Reprod. 2008 Jul;14(7):413-21. doi: 10.1093/molehr/gan029. Epub 2008 Jun 4. PMID 18524812
- [Background] Mirkin S, Arslan M, Churikov D, Corica A, Diaz JI, Williams S, Bocca S, Oehninger S. In search of candidate genes critically expressed in the human endometrium during the window of implantation. Hum Reprod. 2005 Aug;20(8):2104-17. doi: 10.1093/humrep/dei051. Epub 2005 May 5. PMID 15878921
- [Background] Mirkin S, Nikas G, Hsiu JG, Diaz J, Oehninger S. Gene expression profiles and structural/functional features of the peri-implantation endometrium in natural and gonadotropin-stimulated cycles. J Clin Endocrinol Metab. 2004 Nov;89(11):5742-52. doi: 10.1210/jc.2004-0605. PMID 15531538